CLINICAL TRIAL: NCT01312181
Title: HealthCall: Brief Intervention to Reduce Drug Use in HIV Primary Care
Brief Title: HealthCall:Brief Intervention to Reduce Non-injecting Drug Use in HIV Primary Care Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Principal Investigator, Efrat Aharonovich, Resarch Scientist, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DA024606 (NIH)
Record Dates: First submitted 2011-03-09; First posted 2011-03-10 (Estimated); Results first posted 2018-05-15 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Mental and Behavioral Disorders Due to Harmful Drug Use
Keywords: Technology based intervention; HIV primary care clinic; Brief behavioral intervention; Drug abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors blind to randomization outcomes
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HealthCall +Motivational Interviewing (Active Comparator): Patients access HealthCall by calling a toll-free number and putting a four-digit Personal Identification Number (PIN). The HealthCall system will then ask a short script of pre-recorded questions in English or Spanish, on substance use and other variables (e.g., medication adherence, unprotected sex, feeling of physical well-being, stress, etc). The MI session focuses on reduce ambivalence and increase motivation to reduce non-injection drug use (NIDU), gain a commitment to change, if possible, and ultimately to reduce or eliminate NIDU. The intervention includes: a) identifying pros and cons of using and stopping; b) exploring ambivalence about stopping NIDU; c) eliciting change talk
  Interventions: Behavioral: HealthCall and Motivational Interviewing
- Motivational Interviewing (MI) (Active Comparator): The MI session focuses on reduce ambivalence and increase motivation to reduce non-injection drug use (NIDU), gain a commitment to change, if possible, and ultimately to reduce or eliminate NIDU. The intervention includes: a) identifying pros and cons of using and stopping; b) exploring ambivalence about stopping NIDU; c) eliciting change talk
  Interventions: Behavioral: Motivational Interviewing (MI)
- HIV/AIDS health education - DVD control (Placebo Comparator): HIV/AIDS health education - DVD control. The purpose of this condition is to control for clinical attention associated with Motivational Interviewing (MI)participation, and to provide an analogue of standard care, i.e. brief advice but no other intervention.
  Interventions: Behavioral: HIV/AIDS health education

INTERVENTIONS:
Behavioral: HealthCall and Motivational Interviewing — Patients access HealthCall by calling a toll-free number and putting a four-digit Personal Identification Number (PIN). The HealthCall system will then ask a short script of pre-recorded questions in English or Spanish, on substance use and other variables (e.g., medication adherence, unprotected sex, feeling of physical well-being, stress, etc). The MI session focuses on reduce ambivalence and increase motivation to reduce non-injection drug use (NIDU), gain a commitment to change, if possible, and ultimately to reduce or eliminate NIDU. The intervention includes: a) identifying pros and cons of using and stopping; b) exploring ambivalence about stopping NIDU; c) eliciting change talk
  Arms: HealthCall +Motivational Interviewing
Behavioral: Motivational Interviewing (MI) — The MI session focuses on reduce ambivalence and increase motivation to reduce non-injection drug use (NIDU), gain a commitment to change, if possible, and ultimately to reduce or eliminate NIDU. The intervention includes: a) identifying pros and cons of using and stopping; b) exploring ambivalence about stopping NIDU; c) eliciting change talk
  Arms: Motivational Interviewing (MI)
Behavioral: HIV/AIDS health education — The purpose of this condition is to control for clinical attention associated with Motivational Interviewing (MI)participation, and to provide an analogue of standard care, i.e. brief advice but no other intervention.
  Arms: HIV/AIDS health education - DVD control

SUMMARY:
Among HIV-infected individuals, non-injection drug use (NIDU) is associated with poor HIV medication adherence, greater HIV/AIDS risk behaviors, and increasing non-AIDS mortality. Thus reducing NIDU among HIV infected individuals is critical to their survival and to limiting the spread of HIV. We propose to study the efficacy of a technologically enhanced brief intervention (HealthCall) to reduce NIDU in HIV primary care patients that demands little from busy medical staff and is well accepted by patients. In a 3-arm randomized clinical trial will test the efficacy of (a) Motivational Interviewing (MI)+HealthCall; (b) MI-only; and (c) a control condition (advice + DVD HIV health education) in reducing NIDU.

ELIGIBILITY:
Inclusion Criteria:

* All research volunteers will be 18 and older and HIV positive. We will include participants whose primary drug is non-injection use of cocaine, opioids including heroin, or methamphetamines and current use in the past 30 days > 4 days. Participants will need to complete a medically supervised detoxification if such detoxification is required.

Exclusion Criteria:

* Excluded are research volunteers for whom participation would not be clinically appropriate, who clearly could not participate. Psychotic, suicidal or homicidal patients require clinical management that is too intensive for this study, and we have no evidence that MI+HealthCall would be effective among injection drug users. Leaving New York precludes follow-up. Gross psychomotor/cognitive impairments that may hinder patients' HealthCall use. Hearing and severe vision impairments that preclude telephone use precludes randomization to MI+HealthCall.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Efrat Aharonovich, PhD, Principal Investigator — The New York State Psychiatric Institute and Columbia Univeristy
Locations (2):
- United States (2):
  - Mt Sinai Spencer Cox Center for Health, New York, New York
  - Institute for Advanced Medicine, Mt. Sinai services, New York, New York

REFERENCES:
- [Background] Aharonovich E, Greenstein E, O'Leary A, Johnston B, Seol SG, Hasin DS. HealthCall: technology-based extension of motivational interviewing to reduce non-injection drug use in HIV primary care patients - a pilot study. AIDS Care. 2012;24(12):1461-9. doi: 10.1080/09540121.2012.663882. Epub 2012 Mar 20. PMID 22428809
- [Background] Hasin DS, Aharonovich E, O'Leary A, Greenstein E, Pavlicova M, Arunajadai S, Waxman R, Wainberg M, Helzer J, Johnston B. Reducing heavy drinking in HIV primary care: a randomized trial of brief intervention, with and without technological enhancement. Addiction. 2013 Jul;108(7):1230-40. doi: 10.1111/add.12127. Epub 2013 Apr 17. PMID 23432593

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants age > 18 with > 4 days of NIDU during the prior 30 days were recruited from large urban HIV primary care clinics between 2011 and 2014.
Pre-assignment Details: Of 533 individuals assessed, 240 patients were randomized to a treatment condition, and 224 were included in analyses of the results.
Groups:
- HealthCall +Motivational Interviewing: Patients access HealthCall by calling a toll-free number and putting a four-digit Personal Identification Number (PIN). The HealthCall system will then ask a short script of pre-recorded questions in English or Spanish, on substance use and other variables (e.g., medication adherence, unprotected sex, feeling of physical well-being, stress, etc).
  HealthCall and Motivational Interviewing: A basic behavioral intervention used in the 3 arms including the Motivational Interview (MI), the two components of HealthCall (IVR, personalized feedback) and the advice+DVD educational control arm.
- Motivational Interviewing (MI): The MI session focuses on reduce ambivalence and increase motivation to reduce non-injection drug use (NIDU), gain a commitment to change, if possible, and ultimately to reduce or eliminate NIDU. The intervention includes: a) identifying pros and cons of using and stopping; b) exploring ambivalence about stopping NIDU; c) eliciting change talk
  Motivational Interviewing (MI): A basic behavioral intervention used in the 3 arms including the Motivational Interview (MI), the two components of HealthCall (IVR, personalized feedback) and the advice+DVD educational control arm.
- HIV/AIDS Health Education - DVD Control: HIV/AIDS health education - DVD control. The purpose of this condition is to control for clinical attention associated with Motivational Interviewing (MI)participation, and to provide an analogue of standard care, i.e. brief advice but no other intervention.
  HIV/AIDS health education: A basic behavioral intervention used in the 3 arms including the Motivational Interview (MI), the two components of HealthCall (IVR, personalized feedback) and the advice+DVD educational control arm.
Period: Overall Study
Arm/Group | HealthCall +Motivational Interviewing | Motivational Interviewing (MI) | HIV/AIDS Health Education - DVD Control
Started | 80 | 77 | 83
Completed | 78 | 71 | 75
Not Completed | 2 | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HealthCall +Motivational Interviewing | Motivational Interviewing (MI) | HIV/AIDS Health Education - DVD Control | Total
Number analyzed (Participants) | 80 | 77 | 83 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.53 (9.23) | 47.38 (8.31) | 46.72 (10.32) | 46.54 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 15 | 39
  Male | 66 | 67 | 68 | 201
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 23 | 17 | 62
  Not Hispanic or Latino | 58 | 54 | 66 | 178
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 48 | 39 | 45 | 132
  White | 32 | 38 | 38 | 108
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 80 | 77 | 83 | 240

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Days of Primary Drug Used in the Prior 30 Days
Description: One primary study outcome was frequency of drug use, represented by the total number of days of primary drug used in the prior 30 days (NumDU) as derived from the Time Line Follow Back (TLFB).
Time Frame: Assessed at end of treatment (60 days)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | HealthCall +Motivational Interviewing | Motivational Interviewing (MI) | HIV/AIDS Health Education - DVD Control
Number analyzed (Participants) | 78 | 71 | 75
Days | 5.07 (6.7) | 3.61 (5.79) | 4.73 (7.22)

2. Primary Outcome: Total Dollar Value of Primary Drug Used in the Prior 30 Days
Description: One primary study outcome was quantity of drug used in the prior 30 days, represented by the total dollar amount of primary drug used (QuantU) in the prior 30 days, as derived from the Time Line Follow Back (TLFB).
Time Frame: Assessed at end of treatment (60 days)
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | HealthCall +Motivational Interviewing | Motivational Interviewing (MI) | HIV/AIDS Health Education - DVD Control
Number analyzed (Participants) | 78 | 71 | 75
Dollars | 6.70 (9.79) | 6.47 (8.65) | 6.56 (17.04)

ADVERSE EVENTS:
Time Frame: Serious and Other (Not Including Serious) Adverse Events were assessed throughout the data collection period (3 years).
Arm/Group | HealthCall +Motivational Interviewing | Motivational Interviewing (MI) | HIV/AIDS Health Education - DVD Control
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/71 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/71 | 0/75
Other Adverse Events (participants affected / at risk) | 0/78 | 0/71 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No